CLINICAL TRIAL: NCT03036371
Title: Pilot Study of the Impact of Exercise on Hippocampal Behavior
Brief Title: Pilot Study of the Impact of Exercise on Hippocampal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Helen Blair Simpson, Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7418
Record Dates: First submitted 2017-01-03; First posted 2017-01-30 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Anxiety
Keywords: Neurogenesis; Memory; Spatial Processing; Hippocampus; Cognition; Aerobic Exercise
MeSH Terms: conditions — Anxiety Disorders; Spatial Processing | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Intensity Interval Exercise (Experimental): home exercise sessions
  Interventions: Behavioral: High Intensity Interval Exercise

INTERVENTIONS:
Behavioral: High Intensity Interval Exercise — 6 week at-home aerobic exercise protocol

SUMMARY:
The goal of this pilot study is to test the procedural aspects of the behavioral tests and the exercise components of the study. This includes establishing typical scores for anxiety patients in these behavioral tests, and administering and coaching anxiety patients in an at-home exercise regimen. This pilot study will produce the information necessary to design a larger future study including both patients and healthy control participants.

DETAILED DESCRIPTION:
This is a pilot study to explore whether High Intensity Interval Training (HIIT) aerobic exercise can improve performance on hippocampal dependent behaviors or anxiety measures . HIIT is a form of interval training that alternates short periods of high effort exercise with less intense recovery periods. Participants in this study will undertake a 6-week protocol of HIIT exercise, performed at home on a portable stepper device. Outcome measures for this study will be performance on two hippocampus-dependent behaviors and responses to mood and anxiety questionnaires.

The hippocampus is a brain structure that is involved in learning and memory, and is one of the two sites of adult neurogenesis, the process of generating of new neurons from stem cells in the adult mammalian brain. Adult neurogenesis may represent a new target for the treatment of anxiety disorders. The tests in this study consist of a picture-based memory task and a location memory task. Eligible participants will complete both game tasks. In each test, participants will sit in front of a computer and play these games using the computer keyboard or a handheld video game controller.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of Obsessive Compulsive Disorder (OCD), Social Anxiety Disorder (SAD), Generalized Anxiety Disorder (GAD), Panic Disorder (PD), and/or Specific Phobia (SP)
* No use of psychiatric medication in the past 4 weeks (or 8 weeks for fluoxetine)
* Age 18-40
* Ability to tolerate a treatment-free period
* English-speaking
* Body Mass Index (BMI) within normal range
* Willing and able to sign consent form and comply with study procedures

Exclusion Criteria:

* Current or lifetime comorbid psychiatric conditions that significantly elevate the risk of study participation
* Any major medical or neurological problem that might interfere with reliable performance of study tasks or their interpretation, or render participation dangerous
* Pregnant or lactating
* Use of medication that alters the brain
* Clinical symptom severity warranting immediate treatment
* Current rigorous exercise program
* Participation in Cognitive Behavioral Therapy (CBT) psychotherapy for anxiety

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Change in Percent Correct Score for the Treasure Hunt Task (THT) | 6 weeks
  change between baseline and 6 weeks

SECONDARY OUTCOMES:
Change in Percent Correct Score for the Mnemonic Similarity Test (MST) | 6 weeks
  change between baseline and 6 weeks
Change in Depression, Anxiety, and Stress Scale (DASS) | 6 weeks
  change in self-report questionnaire score between baseline and 6 weeks
Change in Intolerance of Uncertainty Scale (IUS) | 6 weeks
  change in self-report questionnaire score between baseline and 6 weeks
Change in Baecke Physical Activity Questionnaire | 6 weeks
  change in self-report questionnaire score between baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helen B Simpson, M.D, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study intended to assess the feasibility of an at-home exercise protocol in a patient population, and to measure within-patient changes from baseline to post-exercise in order to calculate sample sizes needed for a full study. Therefore, the investigators do not plan to share the data of this small pilot study with other researchers.